CLINICAL TRIAL: NCT05360225
Title: Non-interventional Biomarker Study Testing DNA Extracted From Tumour Tissue Biopsy Samples, Using the Therascreen® KRAS RGQ PCR Kit, From Patients With Non-Small Cell Lung Cancer, Screened in Clinical Study (Protocol No. 20190294).
Brief Title: Testing of DNA Extracted From Tumor Tissue Biopsy Samples Using Therascreen KRAS RGQ PCR Kit
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: QMAN-18-0181-1 004
Record Dates: First submitted 2022-04-20; First posted 2022-05-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clinical Performance Study Protocol for therascreen® KRAS RGQ PCR Kit: The KRAS System (extraction kit, analytical kit, instrument and software) will be used to test FFPE biopsy (resected and core needle biopsy [CNB]/fine needle aspiration [FNA]) tumour tissue from NSCLC patients to establish KRAS G12C mutation status. This will be determined using the investigational device at Q2 Solutions Laboratories.
  Interventions: Diagnostic Test: therascreen® KRAS RGQ PCR Kit

INTERVENTIONS:
Diagnostic Test: therascreen® KRAS RGQ PCR Kit — The KRAS Kit is a real-time qualitative PCR assay used on the Rotor-Gene Q MDx instrument for the detection of somatic G12C mutations in the human KRAS oncogene using DNA extracted from formalin fixed paraffin-embedded (FFPE) Non-small Cell Lung Cancer (NSCLC) tissue.

SUMMARY:
A Non-interventional Biomarker Study for the testing of DNA extracted from tumour tissue biopsy samples, using the therascreen® KRAS RGQ PCR Kit, from patients with Non-Small Cell Lung Cancer, screened in Clinical Study (Protocol No. 20190294).

DETAILED DESCRIPTION:
This is a non-interventional, biomarker screening clinical performance study protocol, for the testing of DNA extracted from tumour tissue biopsy samples (resected and core needle biopsy [CNB]/fine needle aspiration [FNA] tumour tissue) obtained from patients with Non-Small Cell Lung Cancer (NSCLC), using the KRAS Kit. A formal hypothesis will not be tested in this study.

Up to 7000 patient tissue samples (from approximately 5000 patients at 500 clinical trial sites), obtained in the Clinical Study (Protocol No. 20190294), will be tested using the KRAS kit. The testing will be performed at the investigational device clinical testing sites, Q2 Solutions Laboratories in the four geographical locations: USA, Singapore, UK and China

ELIGIBILITY:
Inclusion Criteria:

* All patients who provided consent (by signing and dating the ICF for Protocol No.

20190294), may be included in the Clinical Performance Study.

Exclusion Criteria:

* Patients whose tumour tissue biopsy samples that are not Clinical Study Assay evaluable
* Patients with samples identified for the study which have insufficient testing material
* Specimens which have undergone decalcification.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with NSCLC with KRAS G12C mutation positive tumours.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-05-26 (Actual)

PRIMARY OUTCOMES:
patients with NSCLC with KRAS G12C mutation positive tumours. | 5 business days
  To utilize a Clinical Trial Assay, the KRAS Kit, as a screening test in Phase 3 of Clinical Study (Protocol No. 20190294), in order to identify patients with NSCLC with KRAS G12C mutation positive tumours.

CONTACTS AND LOCATIONS:
Locations (1):
- QIAGEN Gaithersburg, Inc, Manchester, United Kingdom